CLINICAL TRIAL: NCT00521365
Title: A Phase IV STudy of the Effectiveness of Quetiapine Extended Release 600mg Once a Day to Control the Symptoms of Manic Phase of Bipolar Disorder.
Brief Title: Effectiveness of Quetiapine XR on the Control of Symptoms of Manic Phase of Bipolar Disorder.
Acronym: EMMY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00017
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-03

CONDITIONS: Bipolar Disorder; Bipolar Affective Psychosis; Mania; Manic Disorder; Manic State
Keywords: Bipolar Disorder; Bipolar Affective Psychosis; Mania; Manic Disorder; Manic State
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Quetiapine Fumarate

ARMS (1):
- Quetapine 600 mg (Experimental)
  Interventions: Drug: Quetiapine 600mg

INTERVENTIONS:
Drug: Quetiapine 600mg — 300 mg quetiapine fumarate tablets for oral use.
  Day 1: One 300 mg tablet in the evening Day 2: Two 300 mg tablet in the evening Day 3 and onwards: Two 300 mg tablets in the evening, efforts must be done to maintain a daily dose of 600 mg/day.

SUMMARY:
The primary purpose of the study is to assess the efficacy of Quetiapine extended release 600mg per day either as monotherapy or combined therapy in the treatment of patients with mania associated to Bipolar disorder. This trial will also assess the life quality and productivity loss improvement for patients from baseline to day 21.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type I Bipolar Disorder in Manic phase according to standard scales and physician criteria.
* Patients of both genders, aged 18-65 years old being at the first episode
* Patients with chronic Bipolar Disorder with at least one previous manic episode 6 months before inclusion, that based on the physician experience are in a manic episode at study entry quality

Exclusion Criteria:

* Psychoactive substance or alcohol abuse or dependence, forbidden medication, pregnancy, rapid cycling patients, intolerance to Quetiapine, clinically severe disease, unstable Diabetes Mellitus, neutropenia, other laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Polanco, MD, Study Director — AstraZeneca Mexico; Doris Gutierrez, MD, Principal Investigator — INP; Julieta Jimenez, Study Chair — AstraZeneca
Locations (7):
- Mexico (7):
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Pedro Garza García, Nuevo León
  - Research Site, San Luis Potosí City, San Luis Potosí
  - Research Site, Mérida, Yucatán
  - Research Site, Durango

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Type I Bipolar Disorder in manic phase with a YMRS (Young Mania Rating Scale) score ≥12 at study entry. Patients of both genders, 18 - 65 years old, with bipolar disorder I according to the Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria.
Groups:
- Quetiapine 600 mg: Once the patient was enrolled, he/she was provided with a bottle that contains enough tablets of quetiapine to complete up-titration regime and whole treatment as follows:
  Day 1: One 300 mg tablet in the evening Day 2: Two 300 mg tablet in the evening Day 3 and onwards: Two 300 mg tablets in the evening, efforts must be done to maintain a daily dose of 600 mg/day.
  This study is a single arm study. All patients received quetiapine XR 600 mg.
Period: Overall Study
Arm/Group | Quetiapine 600 mg
Started | 88 (98 participants were screened and obtain 88 patients who receive study treatment)
Modified Intention to Treat (mITT) | 88 (Participants who have an YMRS assessment at inclusion, and at least one assessment after inclusion)
Per Protocol (PP) Population | 68 (All participants without protocol deviations)
Safety Analysis Set | 88 (All participants who received study treatment)
Completed | 68 (68 participants completed the study and 68 completed without protocol deviations)
Not Completed | 20
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 6
Not completed — Protocol deviation | 2
Not completed — Drug compliance | 3
Not completed — Usage of not allowed drugs | 6

BASELINE CHARACTERISTICS:
Groups:
- Quetiapine 600 mg: Quetiapine Extended release 600 mg per day either as monotherapy or combined therapy
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Age Continuous [Mean (Standard Deviation); unit: Years] — Participants were asked for their age in years at V0
  Years | 36.51 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants] — Participants were classified as male or female during V0.
  Participants
    Female | 53
    Male | 35
Young Mania Rating Scale (YMRS) total score [Mean (Standard Deviation); unit: Scores on a scale] — Young Mania Rating Scale (YMRS) total score at visit 1(day 0). 11 item instrument with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0 = normal; 4 or 8 = most abnormal. Total possible score is 0 - 60.
  Scores on a scale | 32.06 (9.00)
Clinical Global Impression-Severity (CGI-S) total score [Mean (Standard Deviation); unit: Scores on a scale] — Clinical Global Impression-Severity (CGI-S) total score at visit 1( day 0). 1 item instrument with scale range 0 to 7. 0 = patients who were not assessed, 1 = Normal 7 = the most extremely ill patients.
  Scores on a scale | 5.00 (0.80)
European Quality of Life 5 Dimensions (EQ5D) Questionnaire Index [Mean (Standard Deviation); unit: Scores on a scale] — European Quality of Life 5 Dimensions (EQ5D) Total possible score is 0-1 (0 = The worst quality of life; 1 = The best quality of life).
  Scores on a scale | 0.54 (0.3)
European Quality of Life 5 Dimensions (EQ5D) Questionnaire Visual Analogue Scale (VAS) [Mean (Standard Deviation); unit: Scores on a scale] — European Quality of Life 5 Dimensions (Eq5D) Visual Analog Scale (VAS) at visit 1(day 0). European Quality of Life 5 Dimensions (EQ5D) questionnaire part 2 has 1 item with continuous scale range 0 to 100, where 0= the worst quality of life and 100 = the best quality of life.
  Scores on a scale | 55 (27.8)
Safety scales [Mean (Standard Deviation); unit: Scores on a scale] — Simpson-Angus Scale (SAS) and Barnes Akathisia Rating Scale (BARS)total score at visit 1 (day 0). Simpson-Angus Scale (SAS) for evaluating drug-related extrapyramidal syndromes Questionnaire has 6 items with scale range 0 to 3 for each item.0=Normal; 3=Most abnormal. Total possible score is 0-18. Barnes Akathisia Rating Scale (BARS) Questionnaire has 4 items with scale range 0 to 3 for 3 items and 0 to 5 for 1 item. 0=Normal; 3 or 5=Most abnormal. Total possible score is 0-14.
  Scores on a scale
    SAS | 1.12 (2.20)
    BARS | 1.78 (2.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score From Baseline to End of Treatment (Day 21)
Description: Change in the YMRS total score from baseline to Final Visit or Last Observation Carried Forward (LOCF), modified intention to treat (mITT) population. YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0 - 60.
Time Frame: Baseline and 3 weeks
Population: Modified Intention to treat patients (88). Patients who had taken at least one dose of study drug and had at least one evaluable Young Mania Rating Scale at baseline.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | -20.72 (10.2)

2. Secondary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score From Baseline to Visit 2.
Description: Change in the YMRS total score from baseline to visit 2 (1 week) ,. YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0-60.
Time Frame: Baseline and 1 week
Population: Outcome was comparing the data at baseline with the specific data at visit 2(not with the LOCF), since only 78 patients completed YMRS at visit 2 the number of patients analyzed is different respect to the LOCF (88).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 78
Scores on a scale | -11.5 (7.2)

3. Secondary Outcome: Change in the Young Mania Rating Scale (YMRS) Total Score From Baseline to Visit 3
Description: Change in the YMRS total score from baseline to visit 3(2 weeks). YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0-60.
Time Frame: Baseline and 2 weeks
Population: Outcome was comparing the data at baseline with the specific data at visit 3 (not with the LOCF), since only 79 patients completed YMRS at visit 3 the number of patients analyzed is different respect to the LOCF (88).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 79
Scores on a scale | -18.01 (8.2)

4. Secondary Outcome: Number of Participants With Young Mania Rating Scale (YMRS) Response at Final Visit or Last Observation Carried Forward (LOCF)
Description: Number of participants that had Young Mania Rating Scale (YMRS) response at Final Visit or Last Observation Carried Forward (LOCF). A patient is scored as responder if the change from inclusion shows a reduction of 6 points in the YMRS total score.
  YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0 - 60.
Time Frame: 21 days ± 2 days or Last Observation Carried Forward
Measure: Number; unit: Participants
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Participants | 81

5. Secondary Outcome: Number of Participants With Young Mania Rating Scale (YMRS) Remission at Final Visit or Last Observation Carried Forward (LOCF).
Description: Number of participants that had Young Mania Rating Scale (YMRS) remission at Final Visit or Last Observation Carried Forward (LOCF). A patient is classified in remission if his/her final YMRS total score was ≤11.
  YMRS questionnaire has 11 items with scale range 0 to 4 for 7 items and 0 to 8 for 4 items. 0=normal; 4 or 8=most abnormal. Total possible score is 0 - 60.
Time Frame: 21 days ± 2 days or Last Observation Carried Forward
Measure: Number; unit: Participants
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Participants | 49

6. Secondary Outcome: Change in the Clinical Global Impression (CGI) Total Score From Baseline (CGI-S) to Final Visit or Last Observation Carried Forward (LOCF)(CGI-I).
Description: Clinical Global Impression-Severity(CGI-S)is a measurement of illness severity evaluated at baseline. Clinical Global Impression-Improvement(CGI-I)is a measurement of improvement taken at Final Visit (FV) or Last Observation Carried Forward(LOCF).Change CGI Total score is assessed with next equation: CGI-I total score at FV or LOCF - CGI-S score. CGI-S Questionnaire has a scale range 0-7. 0=patients who are not assessed, 1=Normal 7=the most extremely ill patients. CGI-I Questionnaire has a scale range 0-7. 0=patients who are not assessed, 1=Very much improved; 4= No change; 7=Very much worse.
Time Frame: Baseline and 3 weeks
Population: Modified Intention to treat patients mITT- (88), for each outcome measure where mITT is evaluated, population is the group of patients who had taken at least one dose of study drug and had at least one evaluable Young Mania Rating Scale at baseline.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | -3.95 (0.9)

7. Secondary Outcome: Change in the Clinical Global Impression - Improvement (CGI-I) at Final Visit or Last Observation Carried Forward (LOCF).
Description: Change in the CGI- I at Final Visit or Last Observation Carried Forward (LOCF). CGI I Questionnaire has a one item with scale range 0 to 7. 0=patients who ere not assessed, 1=Very much improved; 4= No change; 7=Very much worse.
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | 1.67 (1.2)

8. Secondary Outcome: Change in the Quality of Life Questionnaire EQ5D Index From Baseline to End of the Study.
Description: Total possible index score is 0-1(0=The worsen quality of life; 1=The best Quality of life).
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | 0.31 (0.3)

9. Secondary Outcome: Change in the Quality of Life Questionnaire EQ5D Visual Analogue Scale (VAS) From Baseline to Final Visit or Last Observation Carried Forward (LOCF).
Description: Change from baseline to Final Visit or Last Observation Carried Forward (LOCF). Quality of Life Questionnaire (EQ5D) part 2 has 1 item with continuous scale range 0 to 100. 0=The worsen Quality of Life; 100=The best Quality of life.
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | 27.73 (29.2)

10. Secondary Outcome: Change in the Simpson-Angus Scale (SAS) Total Score From Baseline to Final Visit or Last Observation Carried Forward (LOCF).
Description: Change in the Simpson-Angus Scale (SAS) total score from baseline to Final Visit or Last Observation Carried Forward (LOCF).
  SAS Questionnaire has a 6 items with scale range 0 to 3 for each item.0=Normal; 3=Most abnormal. Total possible score is 0-18.
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | 1.16 (2.2)

11. Secondary Outcome: Change in the Barnes Akathisia Rating Scale (BARS) Total Score From Baseline to Final Visit or Last Observation Carried Forward (LOCF).
Description: Change in the BARS total score from baseline to Final Visit or Last Observation Carried Forward (LOCF). BARS Questionnaire has 4 items with scale range 0 to 3 for 3 items and 0 to 5 for 1 item. 0=Normal; 3 or 5=Most abnormal. Total possible score is 0-14.
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Scores on a scale | 1.78 (2.4)

12. Secondary Outcome: Change in Weight From Baseline to Final Visit or Last Observation Carried Forward (LOCF).
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Kg | 0.27 (1.90)

13. Secondary Outcome: Change in Waist Circumference From Baseline to Final Visit or Last Observation Carried Forward (LOCF).
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
cm | -0.29 (3.90)

14. Secondary Outcome: Number of Participants With >7% Increase in Weight
Description: Number of participants with >7% increase in weight from baseline to end of study.
Time Frame: Baseline and 3 weeks
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Quetiapine 600 mg
Number analyzed (Participants) | 88
Participants | 1

ADVERSE EVENTS:
Arm/Group | Quetiapine 600 mg
Serious Adverse Events (participants affected / at risk) | 1/88
Other Adverse Events (participants affected / at risk) | 30/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine 600 mg (N=88)
Mania Increased (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine 600 mg (N=88)
Akathisia (Nervous system disorders) | 2
Cephalea (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 3
Gastritis (Gastrointestinal disorders) | 2
Hypertriglycerides (Blood and lymphatic system disorders) | 2
Somnolence (Nervous system disorders) | 13
Tachycardia (Vascular disorders) | 2
Tremor (Nervous system disorders) | 2
Anxiety (Nervous system disorders) | 2

LIMITATIONS AND CAVEATS:
Open label, non comparative study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other